CLINICAL TRIAL: NCT05311800
Title: Effect of Two Isoenergetic Modes of High-Intensity Interval Training on Total and Abdominal Fat Mass Loss in Men With Overweight or Obesity.
Brief Title: High-Intensity Interval Training and Fat Mass Losses
Acronym: RIESLING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratoire des Adaptations Métaboliques à l'Exercice en conditions Physiologiques et Pathologiques (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ID-RCB 2019-A02999-48
Record Dates: First submitted 2022-03-16; First posted 2022-04-05 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Overweight and Obesity; Men
Keywords: cycling; running; high-intensity interval training; fat mass; visceral tissue; health
MeSH Terms: conditions — Overweight; Obesity; Multiple Endocrine Neoplasia Type 1 | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: 2 groups : running vs cycling
Who Masked: Participant
Masking Description: Data collected on the volunteers will be made anonymous.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High intensity interval training - BIKE (HIIE BIKE) (Experimental): 10 cycles of speeding up for 45 s at 80-thPHR followed by pedaling slowly (40% thPHR) for 1m30s (37min30s)
  Interventions: Other: Physical activity
- High intensity interval training - RUN (HIIE RUN) (Experimental): 9 cycles of speeding up for 45 s at 80-thPHR followed by pedaling slowly (40% thPHR) for 1m30s (35min15s)
  Interventions: Other: Physical activity

INTERVENTIONS:
Other: Physical activity — Comparison of HIIT mode (running vs cycling)

SUMMARY:
The aims of this study was to compare two isoenergetic HIIT (High-intensity Interval training) programs (cycling vs. running) on body composition, substrate oxidation at rest and during a moderate exercise, muscle functionality, glycaemic control, lipid profile, inflammation, maximal aerobic capacity (VO2max) and gut microbiota composition in men with overweight or obesity.

The investigators hypothesized that both programs could decrease total, abdominal and visceral fat mass but due to differences in muscle solicitation, metabolism adaptation and blood flow, and that running could favors greater fat mass losses.

DETAILED DESCRIPTION:
The first aim of this study was to compare two isoenergetic HIIT programs (cycling vs. running) on body composition in men with overweight or obesity.

20 men with overweight or obesity should completed HIIT program three times a week during twelve weeks.

i) High intensity interval training - BIKE (HIIE BIKE) 10 cycles of speeding up for 45 s at 80-thPHR followed by pedaling slowly (40% thPHR) for 1m30s (37min30s) ii) High intensity interval training - RUN (HIIE RUN) 9 cycles of speeding up for 45 s at 80-thPHR followed by pedaling slowly (40% thPHR) for 1m30s (35min15s)

Body composition will be measured before and after HIIT program by Dual-energy X-ray absorptiometry (DXA).

ELIGIBILITY:
Inclusion Criteria:

* men (18 to 65 years old)
* with overweight or obesity (BMI > 25 kg/m2 and ≤ 40 kg/m2)

Exclusion Criteria:

* medical contraindications to intense physical activity,
* painful joints,
* taking ß-blocker

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
HIIT mode and fat mass change (g) | At the first and the last training - week 1 and 12
  change of total fat mass (in grams from DXA analysis) after 3 months of training- HIIT mode comparison
HIIT mode and abdominal fat mass change (g) | At the first and the last training - week 1 and 12
  change of abdominal fat mass (in grams from DXA analysis) after 3 months of training- HIIT mode comparison

SECONDARY OUTCOMES:
Rate of carbohydrate and lipid oxidation (g.min-1) during a sub-maximal exercise by measuring gaz exchange. | At the first and the last training - week 1 and 12
  Carbohydrate and lipid oxidation rate (g.min-1) during a submaximal exercise before and after the HIIT protocol. HIIT mode comparison.

CONTACTS AND LOCATIONS:
Locations (1):
- CREPS Auvergne Rhône-Alpes / Vichy, Bellerive-sur-Allier, Allier, France

IPD SHARING:
Plan to Share IPD: No